CLINICAL TRIAL: NCT03893513
Title: Comparison of Transthoracic Electrical Bioimpedance and Pulse Contour Analysis in Renal Transplantation Patients: Analysis of Intraoperative Cardiac Output, Systemic Vascular Resistant and Stroke Volume Variation
Brief Title: Comparison of Transthoracic Electrical Bioimpedance and Pulse Contour Analysis in Renal Transplantation Patients
Status: Completed | Type: Observational
Sponsor: Dita Aditianingsih (Other)
Responsible Party: Sponsor-Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: IndonesiaUAnes032
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Hemodynamic Monitoring
Keywords: Bio-impedance; Haemodynamic monitoring; Pulse contour analysis; kidney transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Transthoracic Electrical Bioimpedance — Non-invasive hemodynamic monitor
  Other Names: ICON
Device: Pulse Contour Analysis — Invasive hemodynamic monitor
  Other Names: EV1000

SUMMARY:
Hemodynamics monitoring using non-invasive transthoracic electrical bioimpedance ICON are compatible with standard invasive monitoring using pulse contour analysis EV1000

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 35 kg/m^2

Exclusion Criteria:

* Heart function abnormalities (arrhythmia, AV block, using pacemaker, severe aorta stenosis)
* Morbid obesity
* Bradycardia (< 50 bpm)
* Tachycardia (> 110 bpm)
* refuse to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planned to undergo elective kidney transplantation surgery as recipient
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic correlation | Intraoperative
  Correlation between hemodynamic measured between devices: cardiac index, stroke volume index, systemic vascular resistance index, stroke volume index

SECONDARY OUTCOMES:
Changes in hemodynamic profiles: Cardiac Index | Intraoperative
  The trends of perioperative hemodynamic profiles during and after surgery: cardiac index in L/minutes/m^2
Changes in hemodynamic profiles: Stroke Volume Index | Intraoperative
  The trends of perioperative haemodynamic profiles during and after surgery: stroke volume index in mL/beat/m^2
Changes in hemodynamic profiles: Systemic Vascular Resistance Index | Intraoperative
  The trends of perioperative haemodynamic profiles during and after surgery: systemic vascular resistance index in dynes-second-m^2/cm^5
Changes in hemodynamic profiles: Stroke Volume Variation | Intraoperative
  The trends of perioperative haemodynamic profiles during and after surgery: stroke volume variation in %

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Vincent JL, Pelosi P, Pearse R, Payen D, Perel A, Hoeft A, Romagnoli S, Ranieri VM, Ichai C, Forget P, Della Rocca G, Rhodes A. Perioperative cardiovascular monitoring of high-risk patients: a consensus of 12. Crit Care. 2015 May 8;19(1):224. doi: 10.1186/s13054-015-0932-7. PMID 25953531
- [Background] Joosten A, Huynh T, Suehiro K, Canales C, Cannesson M, Rinehart J. Goal-Directed fluid therapy with closed-loop assistance during moderate risk surgery using noninvasive cardiac output monitoring: A pilot study. Br J Anaesth. 2015 Jun;114(6):886-92. doi: 10.1093/bja/aev002. Epub 2015 Feb 17. PMID 25690834
- [Background] Pearse RM, Harrison DA, MacDonald N, Gillies MA, Blunt M, Ackland G, Grocott MP, Ahern A, Griggs K, Scott R, Hinds C, Rowan K; OPTIMISE Study Group. Effect of a perioperative, cardiac output-guided hemodynamic therapy algorithm on outcomes following major gastrointestinal surgery: a randomized clinical trial and systematic review. JAMA. 2014 Jun 4;311(21):2181-90. doi: 10.1001/jama.2014.5305. PMID 24842135
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Edison E, Pearse R. Goal directed therapy in the perioperative setting: What is the evidence? In: Paradise Lost and the Cosmological Revolution. 2014.
- [Background] Aya HD, Cecconi M, Rhodes A. Perioperative Haemodynamic Optimisation. Turk J Anaesthesiol Reanim. 2014 Apr;42(2):56-65. doi: 10.5152/TJAR.2014.2220141. Epub 2014 Apr 1. PMID 27366392
- [Background] Saugel B, Cecconi M, Wagner JY, Reuter DA. Noninvasive continuous cardiac output monitoring in perioperative and intensive care medicine. Br J Anaesth. 2015 Apr;114(4):562-75. doi: 10.1093/bja/aeu447. Epub 2015 Jan 16. PMID 25596280
- [Background] Alhashemi JA, Cecconi M, Hofer CK. Cardiac output monitoring: an integrative perspective. Crit Care. 2011;15(2):214. doi: 10.1186/cc9996. Epub 2011 Mar 22. No abstract available. PMID 21457508
- [Background] Allaria B, Poli DM CD. Perioperative hemodynamic monitoring: invasive vs. non-invasive. In: Anesthesia, Pain, Intensive Care and Emergency Medicine - APICE. Italy: Springer-Verlag; 2013. p. 291-9.
- [Background] Boyd O, Jackson N. How is risk defined in high-risk surgical patient management? Crit Care. 2005 Aug;9(4):390-6. doi: 10.1186/cc3057. Epub 2005 Feb 9. PMID 16137389
- [Background] Goldfarb D, Poggio E. Etiology, pathogenesis, and management of renal failure. In: Wein A, Kavoussi L, Novick A, Partin A, Peters C, editors. Campbell-Walsh Urology. 10th ed. Philadelphia: Elsevier Saunders; 2012. p. 1226-53.
- [Background] Angelotti T, Lemmens H. Liver/Kidney/Pancreas transplantation. In: Jaffe R, Schmiesing C, Golianu B, editors. Anesthesiologist's Manual of Surgical Procedures. 5th editio. Philadelphia: Wolters Kluwer Health; 2014. p. 1097-100.
- [Background] Darovic G. Hemodynamic monitoring: invasive and noninvasive clinical applications. 3rd ed. Darovic G, editor. Philadelphia: W.B. Saunders; 2002. 191-260 p.
- [Background] Bendjelid K, Marx G, Kiefer N, Simon TP, Geisen M, Hoeft A, Siegenthaler N, Hofer CK. Performance of a new pulse contour method for continuous cardiac output monitoring: validation in critically ill patients. Br J Anaesth. 2013 Oct;111(4):573-9. doi: 10.1093/bja/aet116. Epub 2013 Apr 26. PMID 23625132
- [Background] Kiefer N, Hofer CK, Marx G, Geisen M, Giraud R, Siegenthaler N, Hoeft A, Bendjelid K, Rex S. Clinical validation of a new thermodilution system for the assessment of cardiac output and volumetric parameters. Crit Care. 2012 May 30;16(3):R98. doi: 10.1186/cc11366. PMID 22647561
- [Background] Marque S, Cariou A, Chiche JD, Squara P. Comparison between Flotrac-Vigileo and Bioreactance, a totally noninvasive method for cardiac output monitoring. Crit Care. 2009;13(3):R73. doi: 10.1186/cc7884. Epub 2009 May 19. PMID 19454009
- [Background] Connor C. Commonly used monitoring techniques. In: Barash P, Cullen B, Stoelting R, Cahalan M, Stock C, editors. Clinical Anesthesia. 7th ed. Philadelphia: Lippincott Williams&Wilkins; 2013. p. 712-20.
- [Background] Mehta Y, Arora D. Newer methods of cardiac output monitoring. World J Cardiol. 2014 Sep 26;6(9):1022-9. doi: 10.4330/wjc.v6.i9.1022. PMID 25276302
- [Background] Porhomayon J, El-Solh A, Papadakos P, Nader ND. Cardiac output monitoring devices: an analytic review. Intern Emerg Med. 2012 Apr;7(2):163-71. doi: 10.1007/s11739-011-0738-9. Epub 2011 Dec 7. PMID 22147648
- [Background] Chamos C, Vele L, Hamilton M, Cecconi M. Less invasive methods of advanced hemodynamic monitoring: principles, devices, and their role in the perioperative hemodynamic optimization. Perioper Med (Lond). 2013 Sep 17;2(1):19. doi: 10.1186/2047-0525-2-19. PMID 24472443
- [Background] Peyton PJ, Chong SW. Minimally invasive measurement of cardiac output during surgery and critical care: a meta-analysis of accuracy and precision. Anesthesiology. 2010 Nov;113(5):1220-35. doi: 10.1097/ALN.0b013e3181ee3130. PMID 20881596
- [Background] Frolich M. Cardiovascular monitoring. In: Butterworth J, Mackey D, Wasnick J, editors. Clinical Anesthesiology. 5th ed. New York: McGraw-Hill; 2013. p. 87-122.
- [Background] Suttner S, Schollhorn T, Boldt J, Mayer J, Rohm KD, Lang K, Piper SN. Noninvasive assessment of cardiac output using thoracic electrical bioimpedance in hemodynamically stable and unstable patients after cardiac surgery: a comparison with pulmonary artery thermodilution. Intensive Care Med. 2006 Dec;32(12):2053-8. doi: 10.1007/s00134-006-0409-x. Epub 2006 Oct 13. PMID 17039348 (Retraction: PMID 21604011 Intensive Care Med. 2011 Jul;37(7):1232)
- [Background] Fellahi JL, Caille V, Charron C, Deschamps-Berger PH, Vieillard-Baron A. Noninvasive assessment of cardiac index in healthy volunteers: a comparison between thoracic impedance cardiography and Doppler echocardiography. Anesth Analg. 2009 May;108(5):1553-9. doi: 10.1213/ane.0b013e31819cd97e. PMID 19372335
- [Background] Sodolski T, Kutarski A. Impedance cardiography: A valuable method of evaluating haemodynamic parameters. Cardiol J. 2007;14(2):115-26. PMID 18651447
- [Background] Monnet X, Teboul JL. Minimally invasive monitoring. Crit Care Clin. 2015 Jan;31(1):25-42. doi: 10.1016/j.ccc.2014.08.002. PMID 25435477